CLINICAL TRIAL: NCT03447691
Title: Comparison Between Volatile Anesthetic-desflurane and Total Intravenous Anesthesia With Propofol and Remifentanil on Early Recovery Quality and Long Term Prognosis of Patients Undergoing Pancreatic Cancer and Common Bile Duct Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 4-2017-0662
Record Dates: First submitted 2018-02-11; First posted 2018-02-27 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Pancreatic Cancer or Distal CBD Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Desmin; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * The investigator who research the QoR-40 questionnaire before and after the surgery will not know which group the patient is assigned to.
  * Because of the difference in anesthesia method, it is impossible to apply blindness to an anesthesiologist practicing anesthesia. Thus, the anesthesiologist will maintain anesthesia with the same target in both groups. (anesthesia depth, hemodynamic status and pain control)
  * Blind is released to investigator and outcomes assessor after completion of QoR-40 questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DES Group (Experimental): Desflurane will be administered via tracheal intubation tube at the level of 0.7-1.1 MAC. Remifentanil will be maintained intravenously by continuous infusion rate of 0.01-0.1 mcg / kg / min
  DES Group's anesthetic depth will be adjusted to maintain the BIS (Bispectral index) between 40-60. Vital sign will be maintained within the range of ± 20% of the baseline MBP (Mean BP) and HR (Heart Rate).
  Interventions: Drug: Des (volatile anesthetic-desflurane)
- TIVA Group (Active Comparator): Propofol and remifentanil will be administered via intravenous, using an infusion pump capable of effect site target controlled infusion.
  TIVA Group's anesthetic depth will be adjusted to maintain the BIS (Bispectral index) between 40-60. Vital sign will be maintained within the range of ± 20% of the baseline MBP (Mean BP) and HR (Heart Rate).
  Interventions: Drug: TIVA (Total intravenous anesthesia with propofol and remifentanil)

INTERVENTIONS:
Drug: Des (volatile anesthetic-desflurane) — Inducing unconciouness with 1.5 to 2 mg/kg of propofol, Intubation is performed 3 minutes after administration of remifentanil 1-2 mcg / kg and rocuronium 0.6 mg / kg. Desflurane concentration is maintained 3-7% (0.7-1.1 MAC) and remifentanil continuous infusion (0.02-0.2 mcg / kg / min).
  Arms: DES Group
Drug: TIVA (Total intravenous anesthesia with propofol and remifentanil) — TIVA group is administered with intravenous anesthetic using commercial target controlled infusion (TCI) pump. Anesthesia is induced and maintained with 2-6 mcg / ml propofol and 2-6 ng / ml remifentanil, which are converted to the effect site concentration. After administrating rocuronium 0.6mg/kg, intubation is performed.
  Arms: TIVA Group

SUMMARY:
Investigators asses whether there is any difference in short term recovery and long term prognosis according to the anesthetic method in patients who undergoing pancreatic cancer and bile duct cancer and undergoing surgery for PPPD or distal pancreatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA class I-III who are scheduled to undergo general anesthesia and who are diagnosed with pancreatic cancer or common bile duct cancer and who are scheduled for PPPD or distal pancreatectomy
* patients who voluntarily agree to participate the clinical study after fully informed and understood about the study

Exclusion Criteria:

* there was distant metastasis at the time of diagnosis
* history of drug adverse reaction or use of opioid or sedative drugs before the surgery
* patients who can not communicate enough to answer the survey
* obesity patients over BMI 30
* patient who are expected to maintain ventilator care on the first day of post operation due to the difficult to extubation right after the surgery
* patients who have inappropriate reasons to participate in clinical research

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2017-08-27 (Actual); Primary Completion 2022-08-28 (Estimated); Study Completion 2022-08-28 (Estimated)

PRIMARY OUTCOMES:
score of QoR40 (Quality of Recovery 40) | post operative day #3
  The QoR-40 consists of a total of 40 questionnaires divided into five categories, it is considered to be the most appropriate index to measure the patient's integrated post operation recovery. Our primary outcome is the score of QoR-40 on the third day after surgery

SECONDARY OUTCOMES:
score of QoR40 (Quality of Recovery 40) | post operative day #1
score of QoR40 (Quality of Recovery 40) | post operative day #7

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joe YE, Kang CM, Lee HM, Kim KJ, Hwang HK, Lee JR. Quality of Recovery of Patients Who Underwent Curative Pancreatectomy: Comparison of Total Intravenous Anesthesia Versus Inhalation Anesthesia Using the QOR-40 Questionnaire. World J Surg. 2021 Aug;45(8):2581-2590. doi: 10.1007/s00268-021-06117-0. Epub 2021 Apr 21. PMID 33881579